CLINICAL TRIAL: NCT06512181
Title: Uterine Preservation in the Management of Placenta Accreta Spectrum Disorders
Acronym: U-PRESERVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Beth Pineles, Assistant Professor of Obstetrics and Gynecology,Assistant Professor of Obstetrics and Gynecology in Biostatistics and Epidemiology, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 854957
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Placenta Accreta Spectrum
MeSH Terms: conditions — Placenta Accreta | interventions — Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Uterine preservation (Experimental): Conservative management of PAS with the inclusion of antibiotics and uterine artery embolization, followed by close monitoring.
  Interventions: Other: Conservative/Expectant Management

INTERVENTIONS:
Other: Conservative/Expectant Management — At time of caesarean section, participants will not have a hysterectomy, but will be treated clinically to preserve their uterus.

SUMMARY:
This study for the conservative management of placenta accreta spectrum disorders (PAS), which are a major cause of maternal morbidity and mortality. The most common management strategy for PAS in the United States is a preterm cesarean-hysterectomy. However, accumulating data show that conservative management is safer and is preferred by some patients. In selected participants (n=15) who desire uterine preservation, the investigators provide the option of conservative management, which will be defined as leaving the placenta in the uterus after delivery of the infant. This is a single-arm single-site pilot study where all participants will be carefully monitored during a standard postpartum inpatient stay and with outpatient follow-up until the uterus is empty.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. A person with a uterus, age 18 or older
4. Currently 16-36 weeks pregnant with an intrauterine gestation
5. History of cesarean delivery AND placenta previa OR anterior low-lying placenta AND suspected of having PAS on prenatal imaging (ultrasound/MRI)
6. Patients for whom the usual management would be cesarean-hysterectomy.
7. Patient desires uterine preservation
8. Agreement to adhere to Lifestyle Considerations (see section 5.3) throughout study duration.

Exclusion Criteria:

• Have a low antenatal suspicion for PAS based on imaging.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2030-09-01 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Hysterectomy rate | Delivery through 1 year
  Percent of participants who undergo a hysterectomy

SECONDARY OUTCOMES:
Endometritis rate | Delivery through 1 year
  Percent of participants who have endometritis
Coagulopathy rate | Delivery through 1 year
  Percent of participants who have coagulopathy
Frequency of vaginal bleeding | Delivery through 1 year
  Percent of participants with vaginal bleeding at each time point
Frequency of pelvic pain | Delivery through 1 year
  Percent of participants with pelvic pain at each time point

CONTACTS AND LOCATIONS:
Overall Officials: Beth Pineles, MD PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared given the extremely small sample size and risk of participant identification